CLINICAL TRIAL: NCT04477460
Title: Effect of Thickened Feeds on Clinical Outcomes in Children With Brief Resolved Unexplained Event
Acronym: BRUE
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Daniel Duncan, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: IRB-P00038785; K23DK127251 (NIH)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Brief Resolved Unexplained Event; Apparent Life Threatening Event; Oropharyngeal Dysphagia
MeSH Terms: conditions — Brief, Resolved, Unexplained Event; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with BRUE receiving thickened feeds
  Interventions: Dietary Supplement: Thickened feeds
- Infants with BRUE not receiving thickened feeds
  Interventions: Dietary Supplement: Non-thickened feeds

INTERVENTIONS:
Dietary Supplement: Thickened feeds — Thickened feeds directed by medical team
  Groups: Infants with BRUE receiving thickened feeds
Dietary Supplement: Non-thickened feeds — Non-thickened feeds directed by medical team
  Groups: Infants with BRUE not receiving thickened feeds

SUMMARY:
This observational study will examine the effects of thickened feeds on clinical outcomes and healthcare utilization in infants with brief resolved unexplained event (BRUE).

DETAILED DESCRIPTION:
Brief resolved unexplained events (BRUE) are frightening episodes characterized by the appearance of life-threatening choking, pallor, cyanosis, and limpness in infants. These common events are resource-intensive and current management approaches inadequately address persistent symptoms. Infants with BRUE commonly have oropharyngeal dysphagia with aspiration, which is a modifiable risk factor for persistent symptoms, but there are no studies determining the mechanism behind this swallowing dysfunction and if swallowing interventions reduce morbidity. This is a prospective, longitudinal cohort study of infants who experienced brief resolved unexplained event receiving thickened feedings compared to those not receiving thickened feedings over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Less than 1 year of age
* Admitted to Boston Children's Hospital after experiencing first lifetime brief resolved unexplained event.

Exclusion Criteria:

* Any pre-existing medical diagnoses that exclude brief resolved unexplained event diagnosis including seizure disorders and cyanotic congenital heart disease
* Already receiving thickened liquids for treatment of another condition

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be eligible for the study if they are less than 1 year of age and admitted to Boston Children's Hospital after experiencing first lifetime BRUE
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of persistent symptoms and repeat hospitalizations over 6-month follow-up period | 6 months
  Frequency of persistent symptoms and repeat hospitalizations over the 6 months after enrollment, with a comparison between those receiving and not receiving thickened feeds.

SECONDARY OUTCOMES:
Frequency of persistent symptoms and hospitalization risk over the full 12-month follow-up period | 12 months
  Symptoms and hospitalization risk over the full 12-month follow-up period, optimal period of time needed for thickening, parent-reported anxiety levels, cost of care at Boston Children's Hospital, potential adverse effects of thickening, and urine arsenic levels, all compared between subjects receiving and not receiving thickened feeds.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Duncan, MD, MPH, Principal Investigator — Boston Children's Hospital; Rachel Rosen, MD, MPH, Study Director — Boston Children's Hospital; Sudarshan Jadcherla, MD, Study Director — Nationwide Children's Hospital; Taher Omari, PhD, Study Director — Flinders University; Samuel Nurko, MD, MPH, Study Director — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Duncan DR, Growdon AS, Liu E, Larson K, Gonzalez M, Norris K, Rosen RL. The Impact of the American Academy of Pediatrics Brief Resolved Unexplained Event Guidelines on Gastrointestinal Testing and Prescribing Practices. J Pediatr. 2019 Aug;211:112-119.e4. doi: 10.1016/j.jpeds.2019.04.007. Epub 2019 May 15. PMID 31103259
- [Background] Duncan DR, Amirault J, Mitchell PD, Larson K, Rosen RL. Oropharyngeal Dysphagia Is Strongly Correlated With Apparent Life-Threatening Events. J Pediatr Gastroenterol Nutr. 2017 Aug;65(2):168-172. doi: 10.1097/MPG.0000000000001439. PMID 27741062
- [Background] Duncan DR, Liu E, Growdon AS, Larson K, Rosen RL. A Prospective Study of Brief Resolved Unexplained Events: Risk Factors for Persistent Symptoms. Hosp Pediatr. 2022 Dec 1;12(12):1030-1043. doi: 10.1542/hpeds.2022-006550. PMID 36336644